CLINICAL TRIAL: NCT05239988
Title: National Retrospective Observational Study in Patients Treated With Remdesivir Suffering From SARS-CoV-2 Hospitalized in Internal Medicine
Brief Title: Observational Study in COVID-19 Patients Treated With Remdesivir
Acronym: RECOVER
Status: Completed | Type: Observational
Sponsor: Fadoi Foundation, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: FADOI.02.2021
Record Dates: First submitted 2022-02-09; First posted 2022-02-15 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hospitalization
Keywords: COVID-19 patients; Remdesivir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients treated with Remdesivir: Patients suffering from SARS-CoV-2 and treated with Remdesivir admitted to Internal Medicine Unit
  Interventions: Other: no experimental intervention

INTERVENTIONS:
Other: no experimental intervention — There will not be any experimental intervention. The study will be conducted according with normal clinical practice

SUMMARY:
Taking into account the high number of COVID-19 patients managed in Italian Internal Medicine, Fadoi Foundation (Italian Scientific Society of Internal Medicine) promotes a national retrospective observational study in patients treated with Remdesivir, analyzing the characteristics of patients and their clinical outcome during hospitalization, and thus providing real-life information potentially useful to integrate the evidence produced by studies conducted under experimental conditions and available in the literature.

DETAILED DESCRIPTION:
This is a multicenter observational, retrospective study, which involves the participation of 35 Nationally Representative Internal Medicine Units, for each center data on all patients suffering from SARS-CoV-2 and treated with Remdesivir are expected to be recorded. Each center will have the task of collecting the data of patients hospitalized consecutively proceeding backwards until March 2020.

The study is a no-profit scientific project, promoted by The FADOI Foundation, the Scientific Society of Internal Medicine.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥ 18 years
* diagnosed with radiologically documented SARS-CoV-2 pneumonia
* treated with Remdesivir (according to the criteria defined by AIFA*)
* admitted to Internal Medicine from March 2020 to August 2021.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes all consecutive patients aged ≥ 18 years diagnosed with radiologically documented SARS-CoV-2 pneumonia, treated with Remdesivir (according to the criteria defined by AIFA*) and admitted to Internal Medicine from March 2020 to August 2021.
Sampling Method: Probability Sample
Enrollment: 1004 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
characteristics of COVID-19 patients | 2 months
  describe, under conditions of normal clinical practice ("real-life") the different clinical characteristics of patients suffering from SARS-CoV-2, hospitalized in Internal Medicine and treated with Remdesivir
methods of treatment with Remdesivir and the main outcomes | 2 months
  evaluate the methods of treatment with Remdesivir (initiation of therapy with respect to the onset of symptoms) and the main outcomes (duration of hospitalization, possible clinical worsening, side effects, transfer to Intensive Care, mortality).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Fontanella, MD, Study Director — FADOI FOUNDATION
Locations (30):
- Italy (30):
  - Ospedale "Mons. Giovanni Galliano", Acqui Terme, (AL)
  - Ente Ecclesiastico "F. Miulli", Acquaviva delle Fonti, (BA)
  - Ospedale di Andria, Andria, (BT)
  - P.O. di Garbagnate, Garbagnate Milanese, (MI)
  - Ospedale di Melegnano, Melegnano, (MI)
  - Ospedale Broni-Stradella, Stradella, (PV)
  - P.O. di Polistena, Polistena, (RC)
  - AO "Giuseppe Foscati", Avellino
  - Ospedale "S. Paolo", Bari
  - Ospedale di Bentivoglio, Bologna
  - Ospedale Maggiore di Bologna Medicina D, Bologna
  - P.O. "SS. Trinità", Cagliari
  - Ospedale M. Bufalini di Cesena, Cesena
  - Ospedale di Alba e Bra, Cuneo
  - Ospedale di Faenza, Faenza
  - AOU Careggi, Florence
  - Ospedale "Careggi", Florence
  - P.O di Frattamaggiore, Frattamaggiore
  - Ospedale Galliera, Genova
  - Ospedale del Mare, Napoli
  - Azienda Ospedaliero Universitaria di Novara, Novara
  - A.O.U. di Perugia, Perugia
  - Ospedale di Rimini - Medicina 1 COVID, Rimini
  - Ospedale di Rimini -Sub intensiva COVID, Rimini
  - Ospedale "Vannini", Roma
  - Ospedale Fatebenefratelli Isola Tiberina, Roma
  - PO SS Annunziata AOU Sassari, Sassari
  - Ospedale "San Paolo" di Savona, Savona
  - Ospedale "Mauriziano", Torino
  - Ospedale "Circolo-Macchi", Varese

IPD SHARING:
Plan to Share IPD: No